CLINICAL TRIAL: NCT06983886
Title: The Effect of Local Infiltration of Tranexamic Acid on Postoperative Blood Loss in Orthognathic Surgery : A Randomized Controlled Trial
Brief Title: The Effect of Local Infiltration of Tranexamic Acid on Postoperative Blood Loss in Orthognathic Surgery
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Chanokchon Kongkergkiat, Chanokchon Kongkergkiat, M.D., Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MURA2025/288
Record Dates: First submitted 2025-05-01; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Blood Loss in Patient Undergoing Orthognathic Surgery
Keywords: Postoperative blood loss; Orthognathic surgery; Bilateral sagittal split ramus osteotomies; BSSO; BSSRO; Tranexamic acid
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranexamic Acid; Saline Solution; Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Randomization will be performed using a computer-generated sequence by a research staff member from the Department of Surgery to determine the side of intervention. For example, if the randomized value is 0, the left side will receive the intervention drug and the right side will serve as the control; if the value is 1, the right side will receive the intervention drug and the left side will serve as the control. Block randomization will be used to ensure balanced allocation between the two groups.
  The randomization result will be sealed in an opaque envelope, which will be opened in the operating room prior to surgery by a resident not involved in the surgical procedure. The envelope will contain the randomization assignment and instructions for drug preparation. This uninvolved resident will prepare two syringes labeled for the left (L) and right (R) sides accordingly.
  The randomization assignment will remain blinded to the subject, surgical team, evaluator.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine with adrenaline and normal saline solution (Active Comparator): A local anesthetic solution was prepared by mixing 10 ml of 1% lidocaine with adrenaline (1:100,000) and 5 ml of normal saline (NSS), resulting in a total volume of 15 ml. The solution was injected at the planned mandibular osteotomy sites on both the medial and lateral aspects of the ramus of the mandible. The injection was administered after the induction of general anesthesia, followed by a 5-minute waiting period to allow the anesthetic to take effect before making the surgical incision.
  This solution will be used on either left or right side of mandible depends on the randomized result, and the other side will be given the solution of another arm.
  Interventions: Drug: Normal Saline Solution (NSS); Drug: Lidocaine (drug)
- Lidocaine with adrenaline and tranexamic acid (Experimental): A local anesthetic solution was prepared by mixing 10 ml of 1% lidocaine with adrenaline (1:100,000) and 5 ml of tranexamic acid (50 mg/ml), resulting in a total volume of 15 ml. The solution was injected at the planned mandibular osteotomy sites on both the medial and lateral aspects of the ramus of the mandible. The injection was administered after completion of general anesthesia, followed by a 5-minute waiting period to allow the anesthetic to take effect before the surgical incision was made.
  This solution will be used on either left or right side of mandible depends on the randomized result, and the other side will be given the solution of another arm.
  Interventions: Drug: Tranexamic Acid; Drug: Lidocaine (drug)

INTERVENTIONS:
Drug: Tranexamic Acid — A local anesthetic solution was prepared by mixing 10 ml of 1% lidocaine with adrenaline (1:100,000) and 5 ml of tranexamic acid (50 mg/ml), resulting in a total volume of 15 ml. The solution was injected at the planned mandibular osteotomy sites on both the medial and lateral aspects of the ramus of the mandible. The injection was administered after completion of general anesthesia, followed by a 5-minute waiting period to allow the anesthetic to take effect before the surgical incision was made.
  Arms: Lidocaine with adrenaline and tranexamic acid
Drug: Normal Saline Solution (NSS) — A local anesthetic solution was prepared by mixing 10 ml of 1% lidocaine with adrenaline (1:100,000) and 5 ml of normal saline (NSS), resulting in a total volume of 15 ml. The solution was injected at the planned mandibular osteotomy sites on both the medial and lateral aspects of the ramus of the mandible. The injection was administered after the induction of general anesthesia, followed by a 5-minute waiting period to allow the anesthetic to take effect before making the surgical incision.
  Arms: Lidocaine with adrenaline and normal saline solution
Drug: Lidocaine (drug) — A local anesthetic solution was prepared by mixing 10 ml of 1% lidocaine with adrenaline (1:100,000) and 5 ml of normal saline (NSS) or 5 ml of tranexamic acid (50 mg/ml) depends on allocated group, resulting in a total volume of 15 ml. The solution was injected at the planned mandibular osteotomy sites on both the medial and lateral aspects of the ramus of the mandible. The injection was administered after the induction of general anesthesia, followed by a 5-minute waiting period to allow the anesthetic to take effect before making the surgical incision.

SUMMARY:
The effect of local infiltration of tranexamic acid in orthognathic surgery remains unclear. This study was conducted to evaluate the difference in postoperative blood loss, measured by surgical drain output, following orthognathic surgery. The investigation involved a within-subject comparison, where each side of the mandible received a different local anesthetic solution: one side was infiltrated with a mixture of lidocaine with adrenaline and tranexamic acid, while the other side received lidocaine with adrenaline and normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-50 years
* undergoing orthognathic surgery (Bilateral sagittal split ramus osteotomies (BSSRO), with or without Le Fort I maxillary osteotomy)
* ASA physical status I-II

Exclusion Criteria:

* Genioplasty in the operation
* History of allergy to tranexamic acid
* History of thromboembolic disorders
* Use of medications affecting blood coagulation (antiplatelet or anticoagulants) within the past 2 weeks
* History of cerebrovascular disease
* Pregnant or breastfeeding women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative blood loss | 24 hours and 48 hours after the end of intervention
  Amount of surgical drain output

SECONDARY OUTCOMES:
Postoperative pain score | 24 hours and 48 hours after the end of intervention
  Visual analog scale (0-10) 0 = no pain, 10 = the worst pain
Postoperative edema | At 48 hours and 1 week after the end of intervention
  Standardized frontal facial photographs to determine whether the left side, right side, or both sides were equally swollen. The evaluation was performed by 3 independent assessors.
Surgical filed visibility | Intraoperatively
  Fromme-Boezaart scale 0 = No bleeding (cadaveric conditions)
  1. = Slight bleeding - no suction required
  2. = Slight bleeding - occasional suctioning required
  3. = Slight bleeding - frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed
  4. = Moderate bleeding - frequent suctioning required and bleeding threatens surgical field directly after suction is removed
  5. = Severe bleeding - constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely
Headaches (Adverse events of tranexamic acid) | within one week after end of the intervention
  Patient reported outcome using a questionnaire interview And clinical examination (0=no,1=yes)
Nausea vomiting (Adverse events of tranexamic acid) | within one week after end of the intervention
  Patient reported outcome using a questionnaire interview And clinical examination (0=no,1=yes)
Seizure (Adverse events of tranexamic acid) | within one week after end of the intervention
  Patient reported outcome using a questionnaire interview And clinical examination (0=no,1=yes)
Thromboembolic events (Adverse events of tranexamic acid) | within one week after end of the intervention
  Patient reported outcome using a questionnaire interview And clinical examination (0=none,1=DVT,2=Stroke,3=MI)
Drug allergy (Adverse events of tranexamic acid) | within one week after end of the intervention
  Patient reported outcome using a questionnaire interview And clinical examination (0=no,1=yes : urticaria, MP rash, anaphylaxis)
Local irritation | within one week after end of the intervention
  Patient reported outcome using a questionnaire interview And clinical examination (0=no,1=yes : rash, erythema, itching)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided